CLINICAL TRIAL: NCT06048861
Title: Evaluation of Joint Position Sense With Two Different Electrogoniometers in Mild and Moderate Carpal Tunnel Syndrome
Brief Title: Evaluation of Joint Position Sense in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sinem Yenil, PT, MSc, Research Assistant, Pamukkale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: E-60116787-020-136447
Record Dates: First submitted 2023-09-07; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: joint position sense; electrogoniometer; carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with Carpal Tunnel Syndrome (Experimental)
  Interventions: Device: KForce Sens; Device: Baseline Electrıgoniometer
- Healthy Controls (Experimental)
  Interventions: Device: KForce Sens

INTERVENTIONS:
Device: KForce Sens — The device was attached to the middle of the wrist joint with the help of Velcro for all movements. Starting position of the extremity was determined and this position was introduced to the device as the reference position. Then, the participant was asked to perform the movement.
Device: Baseline Electrıgoniometer — The pivot point of the goniometer was placed next to the ulnar styloid for 30° and 60° wrist flexion and extension, and also it was placed in the middle carpometacarpal joint for radial and ulnar deviation. A passive movement was made to the extremity in a predetermined amount and direction. The participant was asked to remember this position. Then, the participant was asked to return the extremity to this position when their eyes were closed.
  Arms: Individuals with Carpal Tunnel Syndrome

SUMMARY:
The aim of the study was to investigate the validity and reliability of the KForce Sens® for the evaluation of wrist joint position sense in individuals with CTS. Wrist joint position sense was assessed with KForce Sens® and Baseline® electrogoniometer. The validity and reliability of the KForce Sens® for wrist position sense evaluation were investigated by comparing the two data sets.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate CTS confirmed with EMG
* having symptoms for at least 3 months
* not receiving medical treatment and physiotherapy until 3 months before the study at the latest

Exclusion Criteria:

* having trauma in the affected extremity in the last 6 months
* having cervical radiculopathy
* having brachial plexopathy
* having cognitive problems
* having neurological problems
* being pregnant

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Joint position sense | Day 1
  The evaluation of participants' wrist position sense was performed separately with a Baseline® electrogoniometer and KForce Sens®.
Joint position sense re-test | up to 1 week
  The evaluation of participants' wrist position sense was performed with KForce Sens®.

SECONDARY OUTCOMES:
Function and symptom severity | Day 1
  The Boston Carpal Tunnel Questionnaire included 19 items indicating the severity, frequency, and duration of symptoms and difficulty in performing daily tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided